CLINICAL TRIAL: NCT03152422
Title: Urinary Proteomics in Predicting Heart Transplantation Outcomes
Acronym: uPROPHET
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan A. Staessen, Professor of Medicine, KU Leuven
Other Study IDs: ERC PoC 713601-uPROPHET
Record Dates: First submitted 2017-05-08; First posted 2017-05-15 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Urinary proteomics — Urinary proteomics for risk stratification and graft monitoring in recipients of a heart transplant

SUMMARY:
uPROPHET aims to validate urinary proteomics for risk stratification and monitoring graft performance is recipients of heart transplants

DETAILED DESCRIPTION:
The proof of concept underlying uPROPHET rests on the EPLORE findings that capillary electrophoresis coupled with high-resolution mass-spectroscopy reproducibly identified unique urinary proteomic (UP) signatures associated with subclinical left ventricular dysfunction, renal impairment and adverse cardiovascular outcomes. Consensus criteria currently applied for the selection of patients for heart transplantation (HTx) leave an inconvenient margin of uncertainty, because of the unpredictable course of the disease and the shortage of donor hearts. Furthermore, monitoring graft function and adjusting immunosuppression remain major challenges after HTx. Endomyocardial biopsies, up to 20 in the first year after HTx, are the standard approach to detect graft rejection, but require an invasive risk-carrying procedure. uPROPHET aims to develop UP profiling: (1) as a prognostic tool helpful in selecting terminally ill heart failure patients for HTx with the greatest probability of survival while adding a maximum of high-quality years to life; and (2) as an instrument to monitor graft performance and immune system activity and to manage immunosuppression. The new UP classifiers will be initially validated by demonstrating analogy between the proteomic profiles in urine and tissue samples of explanted hearts.

ELIGIBILITY:
Inclusion Criteria:

* End-stage heart failure resistant to treatment

Exclusion Criteria:

* According to guidelines (J Heart Lung Transplant 2010;29:717-27 and J Heart Lung Transplant 2016; 35: http://dx.doi.org/10.1016/j.healun.2015.10.023).

Ages: 10 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: End-stage heart failure due to ischemic, dilated or hypertrophic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular events | Patients were followed up from the date of first urine sampling until death or censoring on the date of the last available follow-up visit (median 4 years). Events will be reported at study completion.
  This endpoint is available in the hospital records

SECONDARY OUTCOMES:
Graft performance | Patients were followed up from the date of first urine sampling until death or censoring on the date of the last available follow-up visit (median 4 years). Events will be reported at study completion.
  Monitoring using endomyocardial biopsies and hemodynamic measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Staessen, MD, PhD, Principal Investigator — University of Leuven

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be made available for scientific purposes via a motivated request to Prof Jan A. Staessen. The request should receive approval by the Ethics Committee of the University Hospitals Leuven.
Supporting Information: Study Protocol, CSR
Time Frame: Currently available until 2025
Access Criteria: Appproval by the Ethics Committee of the University Hospitals Leuven

REFERENCES:
- [Result] Huang QF, Trenson S, Zhang ZY, Yang WY, Van Aelst L, Nkuipou-Kenfack E, Wei FF, Mujaj B, Thijs L, Ciarka A, Zoidakis J, Droogne W, Vlahou A, Janssens S, Vanhaecke J, Van Cleemput J, Staessen JA. Urinary Proteomics in Predicting Heart Transplantation Outcomes (uPROPHET)-Rationale and database description. PLoS One. 2017 Sep 7;12(9):e0184443. doi: 10.1371/journal.pone.0184443. eCollection 2017. PMID 28880921
- [Result] Huang QF, Trenson S, Zhang ZY, Van Keer J, Van Aelst LNL, Yang WY, Nkuipou-Kenfack E, Thijs L, Wei FF, Mujaj B, Ciarka A, Droogne W, Vanhaecke J, Janssens S, Van Cleemput J, Mischak H, Staessen JA. Biomarkers to Assess Right Heart Pressures in Recipients of a Heart Transplant: A Proof-of-Concept Study. Transplant Direct. 2018 Apr 23;4(5):e346. doi: 10.1097/TXD.0000000000000783. eCollection 2018 May. PMID 29796417
- [Result] Huang QF, Zhang ZY, Van Keer J, Trenson S, Nkuipou-Kenfack E, Yang WY, Thijs L, Vanhaecke J, Van Aelst LNL, Van Cleemput J, Janssens S, Verhamme P, Mischak H, Staessen JA. Urinary peptidomic biomarkers of renal function in heart transplant recipients. Nephrol Dial Transplant. 2019 Aug 1;34(8):1336-1343. doi: 10.1093/ndt/gfy185. PMID 29982668
- [Result] Huang QF, Van Keer J, Zhang ZY, Trenson S, Nkuipou-Kenfack E, Van Aelst LNL, Yang WY, Thijs L, Wei FF, Ciarka A, Vanhaecke J, Janssens S, Van Cleemput J, Mischak H, Staessen JA. Urinary proteomic signatures associated with beta-blockade and heart rate in heart transplant recipients. PLoS One. 2018 Sep 24;13(9):e0204439. doi: 10.1371/journal.pone.0204439. eCollection 2018. PMID 30248148
- See also: Description of study at the website of the University of Leuven — https://www.kuleuven.be/english/research/EU/p/horizon2020/es/erc/uprophet